CLINICAL TRIAL: NCT00520078
Title: Clinicopathological and Molecular Correlation of Acrochordon in Relation to Human Papillomavirus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Other Study IDs: 200701034R
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-02

CONDITIONS: Acrochordon; Skin Tag; Soft Fibroma; Human Papillomavirus; HPV

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Acrochordon, or soft fibroma, is a common benign skin tumor which is generally regarded as a sign of cutaneous aging or as a reaction to friction since it occurs in the intertriginous areas. Recent studies have shown the presence of human papillomaviruses, especially the mucosal types, on some of the intertriginous lesions. This study is to analyze the different clinical presentations of acrochordon and correlate them with pathologic and molecular human papillomavirus findings. Further goal is to improve the ability to differentiate acrochordon and its possible prevention and treatment. Also, it may have an implication on the transmission and prevention of cervical carcinoma.

DETAILED DESCRIPTION:
Acrochordon, also called soft fibroma, skin tag or fibroepithelial polyp, is a common cutaneous disorder characterized by a polypoid growth composed of fibroblasts in a loose collagenous stroma, sometimes with proliferation of blood vessels. They appear as soft, skin-colored or light brownish skin tumors. Three types of lesions may occur, (1) multiple small, furrowed papules, especially on the neck and in the axillae, (2) single or multiple filiform smooth growths in various locations, and (3) solitary bag-like pedunculated growth, seen most commonly on the lower trunk. Most regard them as a sign of cutaneous aging.

The presence of human papillomaviruses (HPVs), especially the mucosal types, has been demonstrated in acrochordon. Our previous experience on HPV typing of skin tags also confirms this finding. Though HPV is a ubiquitous virus, the presence of mucosal type HPV in non-mucosal sites is exceptional. This investigation is trying to correlate the clinicopathological and HPV molecular typing of acrochordons. A better understanding of acrochordon and its relation to HPV infection may improve the ability to prevent and treat.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with multiple acrochordon on non-anogenital sites who ask to remove the lesions and have signed consent to surgery will be asked to participate in the study

Exclusion Criteria:

* No special exclusion criteria

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tsen-Fang Tsai, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan